CLINICAL TRIAL: NCT02198794
Title: An Open-Label, Long-Term Safety Study of SD-809 (Deutetrabenazine) for the Treatment of Moderate to Severe Tardive Dyskinesia
Brief Title: Reducing Involuntary Movements in Participants With Tardive Dyskinesia
Acronym: RIM-TD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auspex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SD-809-C-20; 2014-001891-73 (EudraCT Number)
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Tardive Dyskinesia
Keywords: Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms
MeSH Terms: conditions — Tardive Dyskinesia; Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: SD-809 (Experimental): Participants will receive SD-809 orally twice daily (BID) starting at 12 mg/day, which will be titrated based on dyskinesia control and tolerability up to a maximum total dose of 48 mg/day. Participants who decline to participate in Part B, will continue at their stable dose of SD-809 BID up to Week 158.
  Interventions: Drug: SD-809
- Part B: Placebo (Placebo Comparator): Participants will receive placebo matched to SD-809 for 1 week in randomized withdrawal period and thereafter will receive SD-809 (stable dose) for 12 weeks.
  Interventions: Drug: SD-809; Drug: Placebo
- Part B: SD-809 (Active Comparator): Participants will receive SD-809 (stable dose) for 1 week in randomized withdrawal period and will continue to receive the same dose of SD-809 for an additional 12 weeks.
  Interventions: Drug: SD-809
- Part C: SD-809 (Experimental): EU participants who complete Part B and willing to continue in the study will continue treatment with SD-809 for 52 weeks at the dose administered during the 12-week open-label period of Part B.
  Interventions: Drug: SD-809

INTERVENTIONS:
Drug: SD-809 — SD-809 will be administered per dose and schedule specified in the arm.
  Other Names: Deutetrabenazine; TEV-50717
Drug: Placebo — Placebo matching to SD-809 will be administered per schedule specified in the arm.
  Arms: Part B: Placebo

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability, and efficacy of SD-809 in reducing the severity of abnormal involuntary movements of moderate to severe tardive dyskinesia. The purpose of part B is to establish the durability of effect of SD-809 following 1-week period of randomized withdrawal (SD-809 and placebo), followed by 12 weeks of maintenance with SD-809.

DETAILED DESCRIPTION:
Participants who complete study SD-809-C-18 (NCT02195700), SD-809-C-23 (NCT02291861), or any other SD-809 study will be enrolled in this study. This study include a screening period (Part A), a titration period (Part A), a long-term treatment period (Part A), a double-blind, randomized withdrawal period (Part B), treatment after completion of the randomized withdrawal period (Part B), and a post-treatment safety follow-up period (Part A and Part B). EU participants who complete Part B will be invited to participate in Part C.

ELIGIBILITY:
Inclusion Criteria:

* History of using a dopamine receptor antagonist for at least 3 months
* Clinical diagnosis of tardive dyskinesia and has had symptoms for at least 3 months prior to screening
* Participant has successfully completed a controlled study of SD-809 for treatment of moderate to severe tardive dyskinesia
* Participants with underlying psychiatric diagnosis are stable and have no change in psychoactive medications
* Have a mental health provider and does not anticipate any changes to treatment regimen in the next 3 months
* History of being compliant with prescribed medications
* Able to swallow study drug whole
* Be in good general health and is expected to attend all study visits and complete study assessments
* Female participants must not be pregnant and agree to an acceptable method of contraception

Exclusion Criteria:

* Currently receiving medication for the treatment of tardive dyskinesia
* Have a neurological condition other than tardive dyskinesia that may interfere with assessing the severity of dyskinesias
* Have a serious untreated or undertreated psychiatric illness
* Have recent history or presence of violent behavior
* Have unstable or serious medical illness
* Have evidence of hepatic impairment
* Have evidence of renal impairment
* Have known allergy to any component of SD-809 or tetrabenazine
* Has participated in an investigational drug or device trial (other than Study C-18, Study C-23, or any other eligible TEV-50717 parent study) and received study drug within 30 days
* Have acknowledged use of illicit drugs
* Have a history of alcohol or substance abuse in the previous 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, M.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (82):
- United States (44):
  - Teva Investigational Site 145, Tuscaloosa, Alabama
  - Teva Investigational Site 107, Anaheim, California
  - Teva Investigational Site 108, Anaheim, California
  - Teva Investigational Site 123, Glendale, California
  - Teva Investigational Site 160, Irvine, California
  - Teva Investigational Site 176, Loma Linda, California
  - Teva Investigational Site 121, Los Angeles, California
  - Teva Investigational Site 147, Los Angeles, California
  - Teva Investigational Site 174, Norwalk, California
  - Teva Investigational Site 130, Oceanside, California
  - Teva Investigational Site 102, Orange, California
  - Teva Investigational Site 104, San Bernardino, California
  - Teva Investigational Site 110, San Diego, California
  - Teva Investigational Site 169, San Rafael, California
  - Teva Investigational Site 129, Englewood, Colorado
  - Teva Investigational Site 139, New Haven, Connecticut
  - Teva Investigational Site 156, Washington D.C., District of Columbia
  - Teva Investigational Site 157, Boca Raton, Florida
  - Teva Investigational Site 117, Gainesville, Florida
  - Teva Investigational Site 150, Lake City, Florida
  - Teva Investigational Site 153, Miami, Florida
  - Teva Investigational Site 162, Miami, Florida
  - Teva Investigational Site 112, Orlando, Florida
  - Teva Investigational Site 144, Port Charlotte, Florida
  - Teva Investigational Site 155, Augusta, Georgia
  - Teva Investigational Site 165, Decatur, Georgia
  - Teva Investigational Site 131, Chicago, Illinois
  - Teva Investigational Site 154, Baltimore, Maryland
  - Teva Investigational Site 101, Glen Burnie, Maryland
  - Teva Investigational Site 118, Creve Coeur, Missouri
  - Teva Investigational Site 142, Kansas City, Missouri
  - Teva Investigational Site 175, St Louis, Missouri
  - Teva Investigational Site 161, St Louis, Missouri
  - Teva Investigational Site 178, Lincoln, Nebraska
  - Teva Investigational Site 128, Albuquerque, New Mexico
  - Teva Investigational Site 146, Raleigh, North Carolina
  - Teva Investigational Site 114, Garfield Heights, Ohio
  - Teva Investigational Site 133, Charleston, South Carolina
  - Teva Investigational Site 149, Memphis, Tennessee
  - Teva Investigational Site 151, Fort Worth, Texas
  - Teva Investigational Site 115, Salt Lake City, Utah
  - Teva Investigational Site 141, Salt Lake City, Utah
  - Teva Investigational Site 167, Richland, Washington
  - Teva Investigational Site 166, Waukesha, Wisconsin
- Czechia (6):
  - Teva Investigational Site 559, Havířov
  - Teva Investigational Site 556, Hostivice
  - Teva Investigational Site 535, Litoměřice
  - Teva Investigational Site 557, Pilsen
  - Teva Investigational Site 533, Prague
  - Teva Investigational Site 530, Prague
- Germany (2):
  - Teva Investigational Site 502, Gera
  - Teva Investigational Site 504, Mainz
- Hungary (6):
  - Teva Investigational Site 540, Balassagyarmat
  - Teva Investigational Site 538, Budapest
  - Teva Investigational Site 541, Budapest
  - Teva Investigational Site 539, Doba
  - Teva Investigational Site 546, Győr
  - Teva Investigational Site 545, Kalocsa
- Poland (19):
  - Teva Investigational Site 514, Bełchatów
  - Teva Investigational Site 554, Bialystok
  - Teva Investigational Site 510, Bydgoszcz
  - Teva Investigational Site 519, Bydgoszcz
  - Teva Investigational Site 536, Bydgoszcz
  - Teva Investigational Site 523, Chełmno
  - Teva Investigational Site 517, Choroszcz
  - Teva Investigational Site 513, Gdansk
  - Teva Investigational Site 512, Katowice
  - Teva Investigational Site 552, Katowice
  - Teva Investigational Site 520, Krakow
  - Teva Investigational Site 509, Krakow
  - Teva Investigational Site 508, Lodz
  - Teva Investigational Site 511, Lublin
  - Teva Investigational Site 524, Lublin
  - Teva Investigational Site 549, Olsztyn
  - Teva Investigational Site 522, Torun
  - Teva Investigational Site 550, Warsaw
  - Teva Investigational Site 516, Wroclaw
- Slovakia (5):
  - Teva Investigational Site 529, Bratislava
  - Teva Investigational Site 525, Domaša
  - Teva Investigational Site 527, Košice
  - Teva Investigational Site 528, Rimavská Sobota
  - Teva Investigational Site 526, Rožňava

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.)

REFERENCES:
- [Derived] Frank S, Anderson KE, Fernandez HH, Hauser RA, Claassen DO, Stamler D, Factor SA, Jimenez-Shahed J, Barkay H, Wilhelm A, Alexander JK, Chaijale N, Barash S, Savola JM, Gordon MF, Chen M. Safety of Deutetrabenazine for the Treatment of Tardive Dyskinesia and Chorea Associated with Huntington Disease. Neurol Ther. 2024 Jun;13(3):655-675. doi: 10.1007/s40120-024-00600-1. Epub 2024 Apr 1. PMID 38557959
- [Derived] Fernandez HH, Stamler D, Davis MD, Factor SA, Hauser RA, Jimenez-Shahed J, Ondo WG, Jarskog LF, Woods SW, Bega D, LeDoux MS, Shprecher DR, Anderson KE. Long-term safety and efficacy of deutetrabenazine for the treatment of tardive dyskinesia. J Neurol Neurosurg Psychiatry. 2019 Dec;90(12):1317-1323. doi: 10.1136/jnnp-2018-319918. Epub 2019 Jul 10. PMID 31296586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 343 participants who completed previous SD-809 studies, including study SD-809-C-18 (NCT02195700) or SD-809-C-23 (NCT02291861) were enrolled and 337 participants were eligible for analysis. 6 participants were not evaluable and were excluded from the analysis due to site data integrity issues as reported to the United States Food and Drug Administration (US FDA).
Pre-assignment Details: Study included 3 parts: A, B, and C. Participants in Part A who were on a stable dose for ≥4 weeks after a 6-week titration, were invited to participate in Part B. Participants who are noted as "Completed" for Part A: completed the study in Part A plus continued in Part B. EU participants who completed Part B were invited to participate in Part C.
Groups:
- SD-809: Participants received SD-809 orally BID starting at 12 mg/day, which was titrated based on dyskinesia control and tolerability up to a maximum total dose of 48 mg/day. Participants who declined to participate in Part B, continued at their stable dose of SD-809 BID up to Week 158.
- Part B: Placebo: Participants received placebo matched to SD-809 for 1 week in randomized withdrawal period and thereafter received SD-809 (stable dose) for 12 weeks.
- Part B: SD-809: Participants received SD-809 (stable dose) for 1 week in randomized withdrawal period and continued to receive the same dose of SD-809 for an additional 12 weeks.
- Part C: SD-809: EU participants who completed Part B and were willing to continue in the study continued treatment with SD-809 for 52 weeks at the current dose administered during the 12-week open-label period of Part B.
Period: Part A: Open-Label (158 Weeks)
Arm/Group | SD-809 | Part B: Placebo | Part B: SD-809 | Part C: SD-809
Started | 337 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 337 | 0 | 0 | 0
Intent-to-Treat (ITT) Population (All participants who enrolled in the study, regardless of whether or not received study drug.) | 337 | 0 | 0 | 0
Participants Who Participated in Part A But Not in Part B | 195 | 0 | 0 | 0
Participants Who Agreed to Continue in Part B | 142 | 0 | 0 | 0
Completed (Participants who are noted as "Completed" for Part A: completed the study in Part A (Week 158) plus continued in Part B.) | 32 | 0 | 0 | 0
Not Completed | 305 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 79 | 0 | 0 | 0
Not completed — Adverse Event | 33 | 0 | 0 | 0
Not completed — Lost to Follow-up | 24 | 0 | 0 | 0
Not completed — Lack of Efficacy | 9 | 0 | 0 | 0
Not completed — Death | 8 | 0 | 0 | 0
Not completed — Noncompliance with study drug | 3 | 0 | 0 | 0
Not completed — Other than specified | 5 | 0 | 0 | 0
Not completed — Study terminated | 1 | 0 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 0 | 0
Not completed — Agreed to continue in Part B | 142 | 0 | 0 | 0
Period: Part B: Randomized (13 Weeks)
Arm/Group | SD-809 | Part B: Placebo | Part B: SD-809 | Part C: SD-809
Started (Randomized withdrawal ITT population) | 0 | 71 (Participants of Part A who agreed to participate in Part B) | 71 (Participants of Part A who agreed to participate in Part B) | 0
Randomized Withdrawal mITT Population | 0 | 63 | 65 | 0
Completed | 0 | 66 | 68 | 0
Not Completed | 0 | 5 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0
Period: Part C: Safety Assessment (52 Weeks)
Arm/Group | SD-809 | Part B: Placebo | Part B: SD-809 | Part C: SD-809
Started | 0 | 0 | 0 | 80
Completed | 0 | 0 | 0 | 73
Not Completed | 0 | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: ITT population included all participants who were enrolled in the study, regardless of whether or not a participant received a dose of study drug.
Arm/Group | SD-809
Number analyzed (Participants) | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188
  Male | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 300
  Unknown or Not Reported | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 1
  Race: Asian | 2
  Race: Black | 69
  Race: White | 264
  Race: Other | 1
Total Motor Abnormal Involuntary Movement Scale (AIMS) Score [Mean (Standard Deviation); unit: units on a scale] — AIMS is composed of 12 clinician-administered and -scored items. A total motor score from Items 1 to 7 (orofacial, extremity, and truncal movements) was calculated. Items 1 through 7 included facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). Each item was rated on a 5-point anchored scale ranging from 0 (no dyskinesia) to 4 (severe dyskinesia). Total motor AIMS score for Items 1-7 ranged from 0 to 28, with higher scores indicative of more severe dyskinesia.
  units on a scale | 10.7 (4.68)
AIMS Individual Items (8-10) Scores [Mean (Standard Deviation); unit: units on a scale] — AIMS is composed of 12 clinician-administered and -scored items. Item 8 (used as an overall severity index indicating severity of abnormal movements) was rated on a 5-point anchored scale ranging from 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Items 9 and 10 (provide additional information with regard to participant's incapacitation due to abnormal movements and participant's awareness of abnormal movements) were rated on a 5-point anchored scale ranging from 0 (none or no awareness) to 4 (severe or aware, severe distress). Higher scores indicated more severe disease.
  units on a scale
    Severity of abnormal movements | 2.6 (0.78)
    Incapacitation due to abnormal movements | 2.0 (1.07)
    Participant's awareness of abnormal movements | 2.2 (1.08)
Modified Craniocervical Dystonia Questionnaire 24 (CDQ-24) Score [Mean (Standard Deviation); unit: units on a scale] — CDQ-24 is a disease-specific quality of life questionnaire developed for use in participants with craniocervical dystonia. CDQ-24 was modified such that the questions focus more directly on the impact of TD on quality of life. The following domains were evaluated in mCDQ-24: stigma, emotional well-being, pain, activities of daily living, and social/family life. Each of the 24 questions were rated by participants on a scale of 0 = never or no impairment to 4 = always or very severe impairment. Total score ranged from 0 - 96, with higher score indicative of severe impairment.
  units on a scale | 29.2 (18.96)

OUTCOME MEASURES:

1. Primary Outcome: Part A, B, and C: Number of Participants With Treatment-Emergent AEs (TEAEs), Serious TEAEs, Severe TEAEs, Drug-Related TEAEs, and TEAEs Leading to Withdrawal
Description: AEs were analyzed as one group combined for parts A and B per planned analysis. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severe AE=prevents normal daily activities. Drug-related TEAEs: TEAEs with possible, probable, or definite relationship to study drug. Serious AEs: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A treatment-emergent AE was defined as an AE that began after the first administration of study medication or existing AEs that worsened after the first dose of study medication. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to the end of follow-up (4 weeks after the last dose of study drug; mean exposure: up to approximately 866.1 days)
Population: Safety population included all participants who were administered any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SD-809 | Part C: SD-809
Number analyzed (Participants) | 337 | 80
Participants
  Any TEAEs | 269 | 23
  Serious TEAEs | 68 | 5
  Severe TEAEs | 57 | 3
  Drug-Related TEAEs | 154 | 3
  TEAEs Leading to Withdrawal From Study | 42 | 3

2. Primary Outcome: Part B: Change From Day 1 Visit in Total Motor AIMS Score at Day 7 Visit, as Assessed by Blinded Central Video Rating
Description: The AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and -scored items. A total motor score from Items 1 to 7 (orofacial, extremity, and truncal movements) was calculated. Items 1 through 7 included facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). Each item was rated on a 5-point anchored scale ranging from 0 (no dyskinesia) to 4 (severe dyskinesia). Total motor AIMS score for Items 1-7 ranged from 0 to 28, with higher scores indicative of more severe dyskinesia.
Time Frame: Day 1 of Part B, Day 7 of Part B
Population: The randomized withdrawal modified intent-to-treat (mITT) population included all participants enrolled in Part B who received study drug during the randomized withdrawal period and had a total motor AIMS score as assessed by blinded central video rating at both the pre-withdrawal visit and the post-withdrawal visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part B: Placebo | Part B: SD-809
Number analyzed (Participants) | 63 | 65
units on a scale
  Pre-withdrawal | 5.7 (0.55) | 5.0 (0.49)
  Change at Post-withdrawal | 0.6 (0.28) | 0 (0.29)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SD-809; The statistical model was an analysis of covariance (ANCOVA) with treatment group and dopamine receptor antagonist status at the pre-withdrawal visit as fixed effects and the pre-withdrawal visit value as a covariate; Test type: Other; p = 0.121, ANCOVA — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = -0.6, 95% CI 2-sided [-1.42 to 0.17]

3. Secondary Outcome: Part A: Change From Baseline in Total Motor AIMS Score at Week 145, as Assessed by the Site Rating
Description: The AIMS is an assessment tool used to detect and follow the severity of tardive dyskinesia (TD) over time. The AIMS is composed of 12 clinician-administered and -scored items. A total motor score from Items 1 to 7 (orofacial, extremity, and truncal movements) was calculated. Items 1 through 7 included facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). Each item was rated on a 5-point anchored scale ranging from 0 (no dyskinesia) to 4 (severe dyskinesia). Total motor AIMS score for Items 1-7 ranged from 0 to 28, with higher scores indicative of more severe dyskinesia.
Time Frame: Baseline, Week 145
Population: The ITT population included all participants who were enrolled in the study, regardless of whether or not a participant received a dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Part A: SD-809: Participants received SD-809 orally BID starting at 12 mg/day, which was titrated based on dyskinesia control and tolerability up to a maximum total dose of 48 mg/day. Participants who declined to participate in Part B, continued at their stable dose of SD-809 BID up to Week 158.
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 160
units on a scale | -6.6 (0.37)

4. Secondary Outcome: Part A: Change From Baseline in Total Motor AIMS Score at Week 158, as Assessed by the Site Rating
Description: as for outcome 2
Time Frame: Baseline, Week 158
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 34
units on a scale | -6.3 (0.85)

5. Secondary Outcome: Part A: Percent Change From Baseline in Total Motor AIMS Score at Week 145, as Assessed by the Site Rating
Description: as for outcome 2
Time Frame: Baseline, Week 145
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 159
percent change | -57.0 (2.43)

6. Secondary Outcome: Part A: Percent Change From Baseline in Total Motor AIMS Score at Week 158, as Assessed by the Site Rating
Description: as for outcome 2
Time Frame: Baseline, Week 158
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 34
percent change | -54.9 (6.76)

7. Secondary Outcome: Part A: Percentage of Participants Who Had a 50% or Greater Reduction From Baseline in Total Motor AIMS Score, as Assessed by the Site Rating
Description: as for outcome 2
Time Frame: Baseline to Week 145
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 159
percentage of participants | 67

8. Secondary Outcome: Part A: Percentage of Participants Who Had a 70% or Greater Reduction From Baseline in Total Motor AIMS Score, as Assessed by the Site Rating
Description: as for outcome 2
Time Frame: Baseline to Week 145
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 159
percentage of participants | 42

9. Secondary Outcome: Part A: Change From Baseline in AIMS Items 8, 9, and 10 Score at Week 145, as Assessed by the Site Rating
Description: The AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and -scored items. Items 8 to 10 deal with global severity as judged by the examiner, and the participant's awareness of the movements and the distress associated with them. Item 8 (used as an overall severity index indicating severity of abnormal movements) was rated on a 5-point anchored scale ranging from 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Items 9 and 10 (provide additional information with regard to participant's incapacitation due to abnormal movements and participant's awareness of abnormal movements) were rated on a 5-point anchored scale ranging from 0 (none or no awareness) to 4 (severe or aware, severe distress). Higher scores indicated more severe disease.
Time Frame: Baseline, Week 145
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 160
units on a scale
  Severity of abnormal movements | -1.3 (0.07)
  Incapacitation due to abnormal movements | -1.3 (0.08)
  Participant's awareness of abnormal movements | -1.3 (0.09)

10. Secondary Outcome: Part A: Percentage of Participants Who Were a Treatment Success, Based on the Clinical Global Impression of Change (CGIC)
Description: A treatment success was defined as much or very much improved on the CGIC from baseline of this study. The CGIC is a single-item questionnaire that asks the investigator to assess a participant's TD symptoms at specific visits/weeks after initiating therapy. The CGIC uses a 7-point Likert scale, ranging from -3 to +3 (-3 = very much worse, -2 = much worse, -1 = minimally worse, 0 = not changed, 1 = minimally improved, 2 = much improved, 3 = very much improved), to assess overall response to therapy.
Time Frame: Baseline up to Week 145
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 160
percentage of participants | 73

11. Secondary Outcome: Part A: Percentage of Participants Who Were a Treatment Success, Based on the Patient Global Impression of Change (PGIC)
Description: A treatment success was defined as much or very much improved on the PGIC from baseline of this study. The PGIC is single-item questionnaire that asks the participant to assess their TD symptoms at specific visits/weeks after initiating therapy. The PGIC uses a 7-point Likert scale, ranging from -3 to +3 (-3 = very much worse, -2 = much worse, -1 = minimally worse, 0 = not changed, 1 = minimally improved, 2 = much improved, 3 = very much improved), to assess overall response to therapy.
Time Frame: Baseline up to Week 145
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 161
percentage of participants | 63

12. Secondary Outcome: Part A: Change From Baseline in Modified CDQ-24 Score at Week 158
Description: The CDQ-24 is a disease-specific quality of life questionnaire developed for use in participants with craniocervical dystonia, including both cervical dystonia (CD) and blepharospasm (BPS). The CDQ-24 was modified such that the questions focus more directly on the impact of TD (as opposed to CD/BPS) on quality of life. The following domains were evaluated in the mCDQ-24: stigma, emotional well-being, pain, activities of daily living, and social/family life. Each of the 24 questions were rated by participants on a scale of 0 = never or no impairment to 4 = always or very severe impairment. Total score ranged from 0 - 96, with higher score indicative of severe impairment.
Time Frame: Baseline, Week 158
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part A: SD-809
Number analyzed (Participants) | 39
units on a scale | -6.3 (2.61)

ADVERSE EVENTS:
Time Frame: Baseline up to the end of follow-up (4 weeks after the last dose of study drug; mean exposure: up to approximately 866.1 days)
Description: Adverse events were analyzed as one group combined for Parts A and B and as a separate group for Part C per planned analysis.
Groups:
- Part A and Part B Participants: Participants received SD-809 orally BID starting at 12 mg/day, which was titrated based on dyskinesia control and tolerability up to a maximum total dose of 48 mg/day. Participants who declined to participate in Part B, continued at their stable dose of SD-809 BID up to Week 158. Participants who agreed to participate in Part B, received SD-809 or placebo matched to SD-809 for 1 week in randomized withdrawal period and thereafter received SD-809 (stable dose) for 12 weeks.
Arm/Group | Part A and Part B Participants | Part C: SD-809
All-Cause Mortality (participants affected / at risk) | 8/337 | 2/80
Serious Adverse Events (participants affected / at risk) | 68/337 | 5/80
Other Adverse Events (participants affected / at risk) | 172/337 | 5/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A and Part B Participants (N=337) | Part C: SD-809 (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised non-convulsive epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Hypomania (Psychiatric disorders) | 2 (2) | 0 (0)
Mania (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 2 (4) | 0 (0)
Schizophrenia (Psychiatric disorders) | 5 (5) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Schizophrenia, paranoid type (Psychiatric disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A and Part B Participants (N=337) | Part C: SD-809 (N=80)
Diarrhoea (Gastrointestinal disorders) | 27 (32) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (28) | 2 (2)
Urinary tract infection (Infections and infestations) | 31 (56) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 18 (23) | 0 (0)
Weight decreased (Investigations) | 32 (34) | 0 (0)
Dyskinesia (Nervous system disorders) | 22 (29) | 2 (2)
Headache (Nervous system disorders) | 24 (31) | 0 (0)
Somnolence (Nervous system disorders) | 34 (41) | 0 (0)
Anxiety (Psychiatric disorders) | 41 (51) | 0 (0)
Depression (Psychiatric disorders) | 35 (45) | 0 (0)
Hypertension (Vascular disorders) | 23 (25) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT02198794/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT02198794/SAP_001.pdf